CLINICAL TRIAL: NCT00765830
Title: A 28 Week Extension to a 24 Week Multi-center, Randomized, Double-blind Clinical Trial to Evaluate the Safety and Tolerability of Vildagliptin (50 mg qd) Versus Placebo in Patients With Type 2 Diabetes and Moderate or Severe Renal Insufficiency
Brief Title: Safety and Tolerability of Vildagliptin Versus Placebo in Patients With Type 2 Diabetes and Moderate or Severe Renal Insufficiency (28 Week Extension)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237A23137E1
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2; Renal Insufficiency
Keywords: Type 2 diabetes, vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 50mg qd vildagliptin
  Interventions: Drug: vildagliptin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vildagliptin — 50mg qd
  Arms: 1
Drug: Placebo — qd
  Arms: 2

SUMMARY:
This clinical trial is designed to provide additional information on the safety and tolerability of vildagliptin (50 mg once daily (qd)) when used in patients with type 2 diabetes mellitus (T2DM) and moderate or severe renal insufficiency

ELIGIBILITY:
Inclusion Criteria:

* Complete the core study

Exclusion Criteria:

* Did not comply with core study requirements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2008-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability in patients with T2DM and moderate or severe renal insufficiency over 52 weeks of treatment | 52 weeks

SECONDARY OUTCOMES:
To explore the efficacy of vildagliptin (50 mg qd) versus placebo in patients with T2DM and moderate or severe renal insufficiency | 52 weeks

CONTACTS AND LOCATIONS:
Locations (90):
- Argentina (7):
  - Clinica de Fracturas y Ortopedia, Buenos Aires
  - Hospital Teodoro Alvarez, Buenos Aires
  - Instituto de Investigaciones Clinicas de Mar del Plata, Buenos Aires
  - Instituto Medico Especializado IME, Buenos Aires
  - Hospital Juan Ramon Vidal, Corrientes
  - Clinica Reina Fabiola, Córdoba
  - Hospital Zenon J. Santillan, San Miguel de Tucumán
- Australia (5):
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Heidelberg Repatriation Hospital, Heidelberg Heights
  - SA Endocrine Clinical Research, Keswick
  - Keogh Medical Research Institute, Nedlands Perth
  - St Vincent's Hospital (Melb), Victoria
- Canada (8):
  - ERS Endocrine Research Society, Vancouver, British Columbia
  - Health Sciences Centre - Diabetes Research Group, Winnipeg, Manitoba
  - Co Medica Research Network Inc., Courtice, Ontario
  - Ultra Med Inc., Pointe-Claire, Quebec
  - Centre de Recherche de Laval, Laval
  - Private Office (Gottesman), Ontario
  - Hopital Maisonneuve-Rosemont, Québec
  - Health Sciences Centre - Diabetes Research Group, Winnipeg
- Costa Rica (4):
  - Clínica Vía San Juan, Cartago
  - Clínica de Endocrinología y Diabetes, San José
  - Clínica San Agustín, San José
  - Hospital Clínica Bíblica, San José
- Finland (3):
  - Satakunnan Keskussairaala, Pori
  - Mediwest Research Center, Seinäjoki
  - Tampereen lääkärikeskus Oy, Koskiklinikka, Tampere
- France (7):
  - Cabinet du Dr Arnou, Angers
  - Cabinet du Dr Giraud Philippe, Angers
  - Hôpital Docteur Duchenne, Boulogne-sur-Mer
  - Hopital Albert Michallon, Grenoble
  - Cabinet médical, Laval
  - Hopital Dupuytren, Limoges
  - Hopital Edouard Herriot, Lyon
- Germany (18):
  - Zentralklinikum Augsburg, Augsburg
  - Praxis Dr. Maxeiner, Bad Kreuznach
  - Universitaetsklinik Charitè, Berlin
  - Praxis Dr. Fischer, Darmstadt
  - Praxis Dr. Merker, Dormagen
  - Univ.-Klinikum Erlangen, Erlangen
  - Kardiol. Gemeinschaftspraxis PD Dr. Winkelmann, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Friedrich Schiller Universitaet Jena, Jena
  - CRS Clinical Research Services Gmbh, Kiel
  - I. Medizinische Univ.-Klinik, Kiel
  - Praxis Dr. Hennig, Meissen
  - Praxis Dr. Grimm, München
  - Univ.-Klinikum München, Campus Innenstadt, München
  - Praxis Dr. Schoell, Nuremberg
  - Forschungszentrum Ruhr, KliFoCenter GmbH, Witten
  - Universitaetsklinik im Luitpold-Krankenhaus, Würzburg
- India (6):
  - Gujarat Endocrine Centre, Ahmedabad
  - M V Hospital for Diabetes and Diabetic Research Center, Chennai
  - Coimbatore Diabetes Foundation, Coimbatore
  - S.R. Kalla Memorial Gastro & General Hospital, Jaipur
  - Meenakshi Mission Hospital & Research Centre, Madurai
  - Diabetes Clinic & Research Centre, Nagpur
- Norway (2):
  - Storoklinikken, Oslo
  - St. Olavs Hospital, Endokrinologisk seksjon, Trondheim
- Russia (11):
  - City Clinical Hospital #6, Chelyabinsk
  - City Clinical Hospital #1, Moscow
  - City Clinical Hospital No.11, Moscow
  - MSU of Medicine and Dentistry on the base of CityHospital 23, Moscow
  - MSUMD on the base of City Clinical Hospital #67, Moscow
  - City polyclinic # 17, City Diabetic Centre #3, Saint Petersburg
  - Krestovsky Island Medical Institute, Saint Petersburg
  - Saint- Petersburg State Mtchnikov's Medical Academy, Saint Petersburg
  - Saint-Petersburg State Pavlov's Medical University, Saint Petersburg
  - Site Management Organisation of Clinical Trials Centers, Smolensk
  - Tyumen State Medicine Academy, Tyumen
- Spain (14):
  - Clinica Mediterranea de Neurociencias, Alicante
  - Hospital de la Ribera, Alzira
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Centro de Salud Begonte, Begonte
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General de Jerez de La Frontera, Jerez de la Frontera
  - Ciutat Sanitaria I Universitaria de Bellvitge, L'Hospitalet de Llobregat
  - Complejo Universitario de San Carlos, Madrid
  - Hospital de Merida, Mérida
  - Hospital Son Dureta, Palma de Mallorca
  - Consorci Hospitalari Parc Tauli, Sabadell
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela
  - Eap El Remei - Vic, Vic
- Sweden (5):
  - ME3PLUS Clinical Trials, Gothenburg
  - Njurmedicin, Sahlgrenska Univ.sjukhuset, Gothenburg
  - Metabolmottagningen, Lasarettet, Kristianstad, Kristianstad
  - VO Endokrinologi/Diabetologi Universitetssjukhuset, Lund
  - Ladulaas Kliniska Studier, Skene

REFERENCES:
- See also: Results for CLAF237A23137E1 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5924